CLINICAL TRIAL: NCT02910362
Title: Intra-surgical Evaluation of CATS Tonometer Prism and AMO Versus Alcon Phacoemulsification Machines
Brief Title: Intra-surgical Evaluation of CATS Tonometer Prism and Abbott Medical Optics Versus Alcon Phacoemulsification Machines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intuor Technologies, Inc. (Industry)
Collaborators: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-02
Record Dates: First submitted 2016-09-13; First posted 2016-09-22 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Cataract Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcon phacoemulsification equipment (Experimental): cataract surgery performed with the Alcon phacoemulsification equipment
  Interventions: Device: Alcon phacoemulsification equipment
- AMO phacoemulsification equipment (Active Comparator): cataract surgery with the AMO phacoemulsification equipment
  Interventions: Device: AMO phacoemulsification equipment

INTERVENTIONS:
Device: Alcon phacoemulsification equipment — cataract surgery with Alcon phacoemulsification equipment.
  Arms: Alcon phacoemulsification equipment
Device: AMO phacoemulsification equipment — cataract surgery with AMO phacoemulsification equipment.
  Arms: AMO phacoemulsification equipment

SUMMARY:
This study will measure the dynamic real-time intraocular pressure (IOP) in the anterior chamber during standard phacoemulsification surgery.

What is known:

* Fluidics control is determined to be one of the primary drivers of physician decision making in choosing phacoemulsification equipment.
* Active pressure system fluidic control has a perceived and possibly real (based upon recent literature) improvement in intra-cameral IOP stability and reduced pressure fluctuations.
* Improved fluidics can allow for reduced dynamic IOP fluctuations, in-the-bag positioned phaco tip, and intra-cameral fluid flow all of which will likely improve corneal health post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 or greater

  * Bilateral cataracts for which phacoemulsification extraction and posterior IOL implantation has been planned for both eyes
  * Subjects able to give informed consent
  * Nuclear Sclerotic cataract graded 2+ or 3+
  * Naturally dilated pupil size (in dim light) > 4.0 mm (with no dilation medications) for both eyes
  * Preoperative corneal astigmatism of 2.5 D or less
  * Ages between 55 and 80
  * Availability, willingness, and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* • Uncontrolled systemic disease that in the opinion of the Investigator would put the subject's heath at risk

  * Intraoperative complications
  * Subjects with only one functional eye
  * Those with one eye having poor or eccentric fixation
  * Mild or severe cataracts, predominantly posterior subcapsular cataracts
  * High corneal astigmatism (i.e. those eyes displaying an oval contact image)
  * Those with corneal scarring or who have had corneal surgery including corneal laser surgery
  * Microphthalmos
  * Buphthalmos
  * Severe Dry eyes
  * Blepharospasm
  * Nystagmus
  * Keratoconus
  * Any other corneal or conjunctival pathology or infection.
  * Central corneal thickness greater than 0,600 mm or less than 0,500 mm (2 standard deviations about the human mean)
  * Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus, immunocompromised, etc.)
  * Uncontrolled systemic or ocular disease
  * History of ocular trauma or prior ocular surgery
  * Fuchs Dystrophy
  * Subjects who may be expected to require retinal laser treatment or other surgical intervention, including LRI's
  * Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
  * Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 4.0 mm under mesopic/scotopic conditions)
  * Contact lens usage within 6 months for PMMA contacts lenses, 1 month for gas permeable lenses or 1 week for extended-wear and daily-wear soft contact lens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean McCafferty, MD, Principal Investigator — Arizona Eye Consultants
Locations (1):
- Arizona Eye Consultants, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2016 until December 2016,15 patients were enrolled at Arizona Eye Consultants clinic
Pre-assignment Details: Patients were included in the study based upon meeting inclusion criteria and not meeting exclusion criteria. Patients were randomized to either group based upon a random number generator.
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Alcon Phacoemulsification Equipment | AMO Phacoemulsification Equipment
Started | 8; 16 Eyes | 7; 14 Eyes
Completed | 8; 16 Eyes | 7; 14 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: 16 eyes from 8 subjects for Alcon equipment and 14 eyes from 7 subjects for AMO.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcon Phacoemulsification Equipment | AMO Phacoemulsification Equipment | Total
Number analyzed (Participants) | 8 | 7 | 15
Number analyzed (Eyes) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8) | 66 (8) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With Stable IOP
Description: Determine comparative IOP stability between Abbott and Alcon phacoemulsification equipment.
Time Frame: intraoperative
Population: Eyes with stable IOP
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Alcon Phacoemulsification Equipment | AMO Phacoemulsification Equipment
Number analyzed (Participants) | 8 | 7
Number analyzed (Eyes) | 16 | 14
Eyes | 16 | 14

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Alcon Phacoemulsification Equipment | AMO Phacoemulsification Equipment
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
small population size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less